CLINICAL TRIAL: NCT06265714
Title: The IndONEsia ICCU Registry: a Multicenter Cohort of Intensive Cardiovascular Care Units Patients in Indonesia
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dafsah A. Juzar, MD, MD, PhD, FIHA, FAsCC, FESC, FAPSIC, FSCAI, Indonesia University
Other Study IDs: LB.02.01/VII/005/KEP005/2022
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases; Acute Coronary Syndrome; Heart Failure; Heart Disease, Coronary; Infections; Sepsis; Stroke; Shock; Chronic Kidney Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome; Heart Failure; Coronary Disease; Infections; Sepsis; Stroke; Shock; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One ICCU Registry: The cohort was observed receiving all the necessary treatment in the ICCU.

SUMMARY:
Patients in the Intensive Cardiovascular Care Unit (ICCU) often present with cardiovascular disease (CVD) issues accompanied by various non-cardiovascular conditions. However, a widely applicable scoring system to predict patient outcomes in the ICCU is lacking. Therefore, developing and validating scores for predicting ICCU patient outcomes are warranted. The aims of the IndONEsia ICCU (One ICCU) registry include developing an epidemiological registry of ICCU patients and establishing a multicentre research network to analyse patient outcomes.This nationwide multicenter cohort will capture data from patients receiving cardiovascular critical care treatment in 10 Indonesian hospitals with ICCU facilities. Recorded data will encompass demographic characteristics, physical examination findings at hospital and ICCU admission, diagnoses at ICCU admission, therapy, intervention, complications on days 3 and 5 of in-ICCU care, in-hospital outcomes, and 30-day outcomes. The One ICCU is a large, prospective registry describing the care process and advancing clinical knowledge in ICCU patients. It will serve as an investigational platform for predicting the mortality of ICCU patients.

DETAILED DESCRIPTION:
This prospective cohort registry study protocol comprised all consecutive primary medical ICCU admissions across one speciality hospital and nine general hospitals in Indonesia. The participating hospitals include the specialized National Cardiovascular Center Harapan Kita in Jakarta and nine general hospitals: Dr. Sardjito General Hospital in Yogyakarta, Dr. Wahidin Sudirohusodo General Hospital in Makassar, H. Adam Malik General Hospital in Medan, Dr. Saiful Anwar General Hospital in Malang, Dr. M. Djamil General Hospital in Padang, Dr. Iskak General Hospital in Tulungagung, Prof. Ngoerah General Hospital in Denpasar, Prof. Dr. R. D. Kandou General Hospital Manado, and Dr. Kariadi General Hospital Semarang. Each participating hospital will contribute data for all consecutive medical ICCU admissions for a period of 2 years, from 2021 to 2023. The participating hospitals were carefully selected to represent all regions of Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICCU
* Aged 18 years or older
* Provide consent to participate in the study

Exclusion Criteria:

- Postoperative management following cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria of this study include patients aged ≥ 18 years old who consent to participate in the study. We exclude admissions solely for postoperative management following cardiac surgery. Patients willing to participate in this study are followed up on their day three and five of in-ICCU care, their hospital discharge time, and day 30 following the day of their hospital discharge. Patients who were admitted to the ICCU and meet the inclusion criteria will be informed regarding the details of this study. In cases where patients cannot express their consent to participate in this study (e.g., those with loss of consciousness), informed consent may be obtained from the patients' guardians on their behalf.
Sampling Method: Non-Probability Sample
Enrollment: 12950 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Alive | 1 to 30 days
  Patient alive after being treated in ICCU.
Death | 1 to 30 days
  Patient death after being treated in ICCU.
Readmitted to ICCU | 1 to 30 days
  If a patient is readmitted to the ICCU after being transferred to a regular ward.
Rehospitalization | 1 to 30 days
  Readmission to the hospital within 30 days of discharge after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dafsah Juzar, MD, Principal Investigator — Indonesia University
Locations (9):
- Indonesia (9):
  - Prof. dr. I.G.N.G. Ngoerah General Hospital, Denpasar, Bali
  - Dr. Kariadi General Hospital, Semarang, Central Java
  - Dr. Saiful Anwar General Hospital, Malang, East Java
  - Dr. Iskak General Hospital, Tulungagung, East Java
  - Prof. Dr. R. D. Kandou Manado General Hospital, Manado, North Sulawesi
  - Dr. Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi
  - Dr. M. Djamil Padang General Hospital, Padang, West Sumatra
  - National Cardiovacular Center Harapan Kita, Jakarta
  - Sardjito General Hospital, Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metkus TS, Baird-Zars VM, Alfonso CE, Alviar CL, Barnett CF, Barsness GW, Berg DD, Bertic M, Bohula EA, Burke J, Burstein B, Chaudhry SP, Cooper HA, Daniels LB, Fordyce CB, Ghafghazi S, Goldfarb M, Katz JN, Keeley EC, Keller NM, Kenigsberg B, Kontos MC, Kwon Y, Lawler PR, Leibner E, Liu S, Menon V, Miller PE, Newby LK, O'Brien CG, Papolos AI, Pierce MJ, Prasad R, Pisani B, Potter BJ, Roswell RO, Sinha SS, Shah KS, Smith TD, Snell RJ, So D, Solomon MA, Ternus BW, Teuteberg JJ, van Diepen S, Zakaria S, Morrow DA. Critical Care Cardiology Trials Network (CCCTN): a cohort profile. Eur Heart J Qual Care Clin Outcomes. 2022 Oct 26;8(7):703-708. doi: 10.1093/ehjqcco/qcac055. PMID 36029517